CLINICAL TRIAL: NCT06481592
Title: A Phase 2, Multicenter, Open-label Study of Lifileucel (Tumor-infiltrating Lymphocytes [TIL]) in Participants With Previously Treated Advanced Endometrial Cancer.
Brief Title: A Study of Lifileucel (Tumor-infiltrating Lymphocytes) in Adults With Advanced Endometrial Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOV-END-201
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Endometrial Cancer
Keywords: Tumor Infiltrating Lymphocytes; TIL; Endometrial Cancer; Endometrial; Cell Therapy; Cellular Immunotherapy; IL-2; Non-myeloablative lymphodepletion (NMALD)
MeSH Terms: conditions — Endometrial Neoplasms | interventions — lifileucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with Endometrial Cancer (Experimental)
  Interventions: Biological: Lifileucel

INTERVENTIONS:
Biological: Lifileucel — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After lymphodepleting chemotherapy including cyclophosphamide and fludarabine, participant is infused with lifileucel, followed by IL-2.
  Other Names: Tumor-Infiltrating Lymphocytes; TIL

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of the lifileucel regimen in participants with previously treated endometrial cancer.

DETAILED DESCRIPTION:
The study will enroll participants with advanced endometrial cancer who previously received treatment with platinum-based chemotherapy and an anti-programmed cell death protein-1 (PD-1)/programmed death ligand 1 (PD-L1) agent in a recurrent or advanced setting, either sequentially or in combination.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a histologically confirmed diagnosis of endometrial carcinoma. All histologies, including carcinosarcoma, will be allowed. Uterine sarcoma will not be allowed.
2. Participants who have received the following previous therapies:

   * At least 1 but no more than 4 lines of prior systemic therapy with no more than 2 lines of chemotherapy in any setting (ie, neoadjuvant or adjuvant setting as well as for recurrent, metastatic, or primary unresectable disease. .
   * Participants have received platinum-based chemotherapy and anti-PD-1/PD-L1 therapy.
   * Participants who declined platinum-based chemotherapy regimen and/or an anti-PD-1/PD-L1 therapy or were deemed ineligible for such therapies by the investigator may be considered after discussion with the medical monitor.
   * Systemic therapy counting towards lines of therapy includes chemotherapy, targeted therapy, immunotherapy, and antibody drug conjugates, given alone or in combination. Hormonal therapy does not count as a line of therapy.
   * Participants must have either (i) documented radiographic disease progression during or after the last line of therapy or (ii) discontinued their last line of therapy because of treatment intolerance or toxicity or (iii) with medical monitor discussion, participant/physician decision in the context of stable disease with evidence of tumor growth.
3. Participants who have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and estimated life expectancy of >6 months.
4. Participants having at least one resectable lesion and at least one measurable lesion, following resection of the lesion for TIL generation.
5. Participants who have adequate organ function, including adequate cardiopulmonary function.
6. Participants of childbearing potential must be willing to practice an approved method of highly effective birth control during treatment and up to 12 months after the last dose of study intervention.
7. Participants who are >70 years of age may be allowed to enroll after the investigator discusses with the medical monitor.

Exclusion Criteria:

1. Participants who have symptomatic untreated brain metastases.
2. Participants who have had a history of allogeneic organ transplant or any form of cell therapy involving prior conditioning chemotherapy within the past 20 years.
3. Participants who require systemic steroid therapy > 10 mg/day prednisone or another steroid equivalent dose.
4. Participants who have any form of primary immunodeficiency.
5. Participants who have another primary malignancy within the previous 3 years.
6. Participants who have received or will receive a live or attenuated vaccination within 28 days prior to the start of the NMALD.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 5 Years
  To evaluate the proportion of participants who have a confirmed complete response (CR) or partial response (PR) per RECIST v1.1.

SECONDARY OUTCOMES:
Complete Response Rate | Up to 5 Years
  To evaluate the proportion of participants who have a confirmed complete response (CR) per RECIST v1.1.
Duration of Response | Up to 5 Years
  To measure from the first time that criteria are met for complete response (CR) or partial response (PR) per RECIST v1.1.
Disease Control Rate | Up to 5 Years
  To measure by the percentage of participants with best overall confirmed response of complete response (CR) or partial response (PR) at any time or stable disease (SD) for at least 4 weeks per RICIST v1.1.
Progression-Free Survival | Up to 5 Years
  To evaluate the time from the date of the lifileucel infusion until disease progression per RECIST v1.1.
Overall Survival | Up to 5 Years
  To measure the time from the date of lifileucel infusion to death due to any cause.
Adverse Events | Up to 5 Years
  To characterize the safety and tolerability profile of lifileucel in participants with advanced endometrial cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Iovance Biotherapeutics Study Team, Study Director — Iovance Biotherapeutics
Locations (12):
- United States (12):
  - Honor Health, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - Orlando Health, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Inc., Tampa, Florida
  - Augusta University, Augusta, Georgia
  - UofL Health - Brown Cancer Center, Louisville, Kentucky
  - Barbara Ann Karmanos Cancer Hospital, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Allegheny Health, Pittsburgh, Pennsylvania
  - Avera Medical Group Oncology, Sioux Falls, South Dakota
  - MD Anderson Cancer Center - U of Texas, Houston, Texas